CLINICAL TRIAL: NCT01824784
Title: TopQ Cut-off Determination Study
Status: Completed | Type: Observational
Sponsor: Topcon Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Organization: Topcon Corporation (Industry)
Other Study IDs: DC-03273
Record Dates: First submitted 2013-04-02; First posted 2013-04-05 (Estimated); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Healthy
Keywords: Normal Eyes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To determine optimal cut-off value for TopQ cut-off.

ELIGIBILITY:
Inclusion Criteria:

* No known ocular pathologies

Exclusion Criteria:

* Any known ocular pathologies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sujects that have no known ocular pathologies
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-02; Primary Completion 2013-06 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Retinal Thickness | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sinai, PhD, Principal Investigator — Director of Clinical Marketing
Locations (1):
- Topcon Medical Systems, Inc., Oakland, New Jersey, United States